CLINICAL TRIAL: NCT00167284
Title: Patient Provider Partnership: Improving Diabetes Care in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: UPMC Office of Community Initiatives (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 010157
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes
Keywords: chronic care model, diabetes, community, diabetes education
MeSH Terms: conditions — Diabetes Mellitus | interventions — Physicians; Patient Education as Topic

INTERVENTIONS:
Behavioral: physician and patient education; physician practice redesign

SUMMARY:
With the advent of managed care, increasing responsibility for the care of patients with diabetes is being placed on primary care physicians. Evidence exists that physicians are not meeting established practice guidelines, and outcomes in patients with diabetes are less than optimal. It is thus the objective of this study to institute a community-based diabetes education intervention for both physicians and patients to enhance adherence to guidelines and improve patient outcomes.

We will conduct a chart review (submitted under a separate IRB: #000733) in primary care practices to determine health status and guideline adherence. Following the chart review, physician practices will be assigned to one of three groups: physician + patient education, physician education alone, and usual care. Following the intervention, a repeat chart review will be conducted. Pre and posttest comparisons will be conducted to examine changes primarily in glycemic control, quality of life, patient knowledge, and physician adherence to practice guidelines. Secondarily, we will examine changes in therapeutic intervention, body mass index, and barriers to diabetes care. We will also examine individual barriers to diabetes care and their influence on outcomes in this population. The last phase of the study will encompass a second follow-up visit in which we will examine behavioral factors related to clinical change and sustainability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* over age 18, diagnosed diabetes, physician is participating in study

Exclusion Criteria:

* pregnancy, imprisonment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2001-10; Study Completion 2005-02

PRIMARY OUTCOMES:
A1c
Blood Pressure
Lipids

SECONDARY OUTCOMES:
Quality of Well Being
Empowerment
Physician attitudes
Patient and physician barriers to diabetes care

CONTACTS AND LOCATIONS:
Overall Officials: Janice C Zgibor, PhD, Principal Investigator — University of Pittsburgh